CLINICAL TRIAL: NCT05661487
Title: Correlation MRI - Paraclinical Examination in Sudden Deafness Associated With Vertigo
Acronym: SBAV
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8265
Record Dates: First submitted 2022-12-14; First posted 2022-12-22 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2022-12

CONDITIONS: Vertigo Labyrinthine
Keywords: Vertigo Labyrinthine; Labyrinthitis; Sudden Deafness; Cochlear Diseases
MeSH Terms: conditions — Labyrinthitis; Hearing Loss, Sudden; Cochlear Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute cochleo-vestibular syndrome or labyrinthitis is characterized clinically by the sudden appearance of a great rotatory vertigo and a unilateral sensorineural hearing loss. In this clinical context, MRI is the examination to eliminate differential diagnoses and to make a positive diagnosis of labyrinthitis (supposedly infectious, immunologic or ischemic). The etiologies described are ischemic, infectious or autoimmune, so the risk factors are very variable (cardiovascular, autoimmune or infectious).

Labyrinthitis has been little studied as a clinical entity in its own right. Indeed, studies mainly focus on sudden deafness with subgroups of patients with vertigo.

The incidence of sudden deafness is of the order of 5 to 20 per 100,000 people per year but is probably under-diagnosed.

The individual and medico-economic consequences are similar to those of hearing loss, with an increased risk of dementia, depression, premature death and an increase in health care consumption.

DETAILED DESCRIPTION:
The objective of the study is to evaluate the performance of MRI (sensitivity and specificity) to localize labyrinthine damage in the presence of an acute cochleovestibular syndrome (presumed to be infectious, ischemic or immunologic) compared to the reference paraclinical examinations for each of the structures.

ELIGIBILITY:
Inclusion criteria:

* Patient of legal age (≥18 years)
* MRI diagnosis of labyrinthitis (presumed to be viral, immunologic, or ischemic in origin) at the University Hospitals (HUS) of Strasbourg between 01/01/2014 and 04/30/2021
* Patient with abrupt deafness (a 30 dB drop in hearing thresholds on at least 3 contiguous frequencies for at least 72 hours) associated with unilateral grand rotatory vertigo of abrupt onset
* Patient with severe unilateral acute onset rotary vertigo with acute unilateral hypoacusis.
* Subject who did not express his opposition, after information, to the reuse of his data for the purpose of this research.

Exclusion criteria:

* Subject who expressed opposition to participating in the study.
* History of chronic vertigo,
* Chronic dizziness,
* Presence of a differential diagnosis on MRI (intra-labyrinthine shwannoma, intra-labyrinthine hemorrhage or complicated cholestatoma)
* History of surgery on the inner or middle ear.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Aadult patient with MRI diagnosis of labyrinthitis (presumed to be viral, immunologic, or ischemic in origin) at HUS between 01/01/2014 and 04/30/2021
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2021-08-19 (Actual); Study Completion 2021-09-19 (Actual)

PRIMARY OUTCOMES:
To evaluate the performance of MRI (sensitivity and specificity) to localize labyrinthine damage in the presence of an acute cochleovestibular syndrome | Files analysed retrospectively from from January 01, 2014 to May 30, 2021 will be examined
  The evaluation criterion is the diagnostic performance (sensitivity/specificity) of MRI for each of the structures (basal turn of the cochlea/ 2nd turn of the spire/ 3 semicircular canals, utricle and saccule) in acute labyrinthitis compared to the complementary examinations (Audiogram, VNG, VHIT, cvEMP and VVS)

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'ORL et de Chirurgie Cervico-Faciale - CHU de Strasbourg - France, Strasbourg, France